CLINICAL TRIAL: NCT06639009
Title: To Determine and Compare the Adjunctive Effect of Photobiomodulation With 940nm Diode Laser on Maximal Interincisal Mouth Opening Versus Conventional Non-invasive Management in Moderate Oral Submucous Fibrosis: A Patient and Outcome Assessor Blinded, Multiple- Arm, Randomized, Placebo Controlled Clinical Trial
Brief Title: Effect of Laser Photobiomodulation in Improving Mouth Opening in Oral Submucous Fibrosis
Acronym: OSMFPBMT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Shalini Gupta (Other)
Responsible Party: Sponsor-Investigator, Dr. Shalini Gupta, Additional Professor, All India Institute of Medical Sciences
Organization: All India Institute of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIIMSA2382; AIIMS A2382 (Other: All India Institute of Medical Sciences New Delhi)
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Oral Submucous Fibrosis
Keywords: Oral Submucous Fibrosis; trismus; Burning pain; diode laser; Photobiology; Electromyography; molecular biology; oral health
MeSH Terms: conditions — Oral Submucous Fibrosis; Trismus; Pain

STUDY DESIGN:
Intervention Model Description: A patient and outcome assessor blinded, multiple- arm, randomized, placebo controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The subjects will be blinded to the group assignment as they will receive PBMT ( Active or Sham as per group assignment ) both intraorally and extraorally The outcome assessor will be blinded to the group assignment of the subjects as they will be identified by unique randomization code only
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Sham Comparator): Photobiomodulation therapy given intraorally on bilateral buccal mucosa and extraorally (sham) with conventional non-invasive management.
  Interventions: Other: 940nm diode laser photobiomodulation; Other: Conventional non -Invasive management in Oral Submucous fibrosis
- Group B (Active Comparator): Photobiomodulation therapy given intraorally (bilateral buccal mucosa) and extraorally (bilateral masseter muscle) with conventional non-invasive management.
  Interventions: Other: 940nm diode laser photobiomodulation; Other: Conventional non -Invasive management in Oral Submucous fibrosis
- Group C (Sham Comparator): Sham (Use of laser handpiece with only red guide light and without using the foot pedal which activates the laser)Photobiomodulation therapy(Placebo) (Intraoral and Extraoral) with conventional non-invasive management.
  Interventions: Other: Conventional non -Invasive management in Oral Submucous fibrosis

INTERVENTIONS:
Other: 940nm diode laser photobiomodulation — The surgical handpiece (diameter 0.6cm) will be used without the fibre optic tips in defocused mode and head sanitized before therapy.
  Peak Power : 0.3Watts Power density: 1 Watt/cm2 Fluence: 4J/cm2 per cycle Spot size : 0.28cm2 Distance : 2mm from surface Mode: Continuous, Non- contact mode, circular motion, overlapping, in clockwise concentric manner with laser handpiece perpendicular to surface Duration of cycle : 25 seconds with interval of 30 seconds alternating with other side Cycles per sitting: Four for each side Four Sittings: Day 0,3, 7, and 15 Area of intervention: Bilateral buccal mucosa and masseter muscle Total treatment time per day: 430 seconds/ approx 7 minutes Total treatment time for 4 sittings: approx 28 minutes
  Arms: Group A; Group B
Other: Conventional non -Invasive management in Oral Submucous fibrosis — Brief behavioral Tobacco, areca nut and alcohol habit cessation counseling as per WHO 5As and 5Rs technique at baseline and each follow up.
  Oral prophylaxis Removal of oral irritational factors like sharp teeth, appliances or prosthesis, impacted buccoverted third molars, parafunctional habits Oral hygiene maintenance instructions Oral physiotherapy Control of systemic conditions Removal of all predisposing factors for oral candida infection Advocacy for safe sexual practices Nutrition and diet counseling( seasonal and regional food rich in nutrients, vitamins, antioxidants avoidance of spicy /sour/ hot foods and drinks) Regular surveillance for malignant transformation

SUMMARY:
This a patient and outcome assessor blinded, multiple arm, randomized placebo controlled clinical trial.

The goal of the study is to study the adjunctive effect of 940nm laser photobiomodulation therapy (PBMT) in precancerous condition like moderate Oral submucous Fibrosis in increasing the mouth opening. It will also assess the the effect of PBMT on oral burning sensation cheek flexibility, electromyography of bilateral masseter muscle, inflammatory and fibrogenic cytokines and oral health quality of life at baseline and after 1 and 3 months of PBMT.

Adult subjects fulfilling the selection criteria will be prospectively recruited after ethical clearance and informed written consent. They will be randomized into 3 groups in 1:1 :1 distribution

The three groups are as follows:

Group A: Photobiomodulation therapy given intraorally on bilateral buccal mucosa and extraorally (sham) with conventional non-invasive management.

Group B: Photobiomodulation therapy given intraorally (bilateral buccal mucosa) and extraorally (bilateral masseter muscle) with conventional non-invasive management.

Group C: Sham (Use of laser handpiece with only red guide light and without using the foot pedal which activates the laser)Photobiomodulation therapy(Placebo) (Intraoral and Extraoral) with conventional non-invasive management.

The conventional non invasive management in Oral submucous fibrosis which all the groups will receive are as follows:

Brief behavioral Tobacco, areca nut and alcohol habit cessation counseling as per WHO 5As and 5Rs technique at baseline and each follow up.

Oral prophylaxis Removal of oral irritational factors like sharp teeth, appliances or prosthesis, impacted buccoverted third molars, parafunctional habits Oral hygiene maintenance instructions Oral physiotherapy(Mouth opening and cheek ballooning exercises) Control of systemic conditions (Anemia, Diabetes, hypertension, thyroid disorders) by specialist referral Removal of all predisposing factors for oral candida infection Advocacy for safe sexual practices Nutrition and diet counseling( seasonal and regional food rich in nutrients, vitamins, antioxidants avoidance of spicy /sour/ hot foods and drinks) Regular surveillance for malignant transformation All the outcome parameters will be assessed at baseline and 1 and 3 months after PBMT.

DETAILED DESCRIPTION:
Study design:

A patient and outcome assessor blinded, multiple- arm, randomized, placebo controlled clinical trial Setting: All India Institute of Medical sciences New Delhi

Selection of patients:

Consecutive patients diagnosed with Oral Submucous Fibrosis based on WHO clinical criteria (Warnakulsurya et al 2007, 2021) and classified as Moderate Oral Submucous Fibrosis based on functional staging of More et al 2011 (Functional staging M2 and M3: maximal interincisal distance 15-35 mm) will be prospectively recruited after ethical clearance and informed written consent.

Clinicopathologic characteristics:

The clinical demographics, Tobacco and Areca nut habit history ( Type, quantity, frequency, duration), association with other habits like smoking/ smokeless tobacco with/ without slaked lime, alcohol and addictive drugs will be recorded. The clinical characteristics and staging/grading of OSMF would be recorded as per prepared proforma and protocol. The clinical grading of moderate OSMF will be done according to WHO clinical criteria and More et al 2011 classification. Biopsy of any suspicious oral lesions if found will be done to rule out malignancy and referred to the cancer center for further management and excluded from study. Enrolment of subjects fulfilling the inclusion and none of the exclusion criteria will be done after information and written informed consent before any further investigation. Routine blood investigations to rule out common systemic conditions ( CBC, Blood glucose, LFT, KFT) Participants will be randomized into three arms (1:1:1) Group A: Photobiomodulation therapy (parameters defined below) given intraorally on bilateral buccal mucosa and extraorally (sham) with conventional non-invasive management.

Group B: Photobiomodulation therapy (parameters defined below) given intraorally (bilateral buccal mucosa) and extraorally (bilateral masseter muscle) with conventional non-invasive management.

Group C: Sham (Use of laser handpiece with only red guide light and without using the foot pedal which activates the laser)Photobiomodulation therapy(Placebo) (Intraoral and Extraoral) with conventional non-invasive management.

Randomization:

Block randomization with varying block size will be done using computer generated random numbers using the Nquery software.

Allocation concealment:

Participants will be randomized using sequentially numbered, opaque sealed envelopes (SNOSE). 315 white envelopes will be prepared with aluminum foil sheet and carbon sheet in each. Assigned treatment protocol will be mentioned clearly on a paper and put in each envelope. For each treatment protocol 105 envelopes will be prepared and sealed. Each envelope will have an identifier of trial on its front. Envelopes will be opened sequentially by an operator blinded to the study protocol after which patients will be allotted a study arm as per the treatment mentioned in the envelope. Before opening the envelope we will write the patient's study identifier number, date and operator's signature in front of the envelope, which will be transferred on white paper through carbon paper. Used envelopes will be stored separately until the completion of trial.

Blinding:

The subjects will be blinded to the group assignment as they will receive PBM ( Active or Sham as per group assignment ) both intraorally and extraorally The outcome assessor will be blinded to the group assignment of the subjects as they will be identified by unique randomization code only

Conventional non-invasive management (Usual care):

All subjects in the three groups will receive the same standard conventional non- invasive management advised for moderate OSMF as per current scientific evidence.

Brief behavioral Tobacco, areca nut and alcohol habit cessation counseling as per WHO 5As and 5Rs technique at baseline and each follow up.

Oral prophylaxis Removal of oral irritational factors like sharp teeth, appliances or prosthesis, impacted buccoverted third molars, parafunctional habits Oral hygiene maintenance instructions Oral physiotherapy(Mouth opening and cheek ballooning exercises) Control of systemic conditions (Anemia, Diabetes, hypertension, thyroid disorders) by specialist referral Removal of all predisposing factors for oral candida infection Advocacy for safe sexual practices Nutrition and diet counseling( seasonal and regional food rich in nutrients, vitamins, antioxidants avoidance of spicy /sour/ hot foods and drinks) Regular surveillance for malignant transformation

Photobiomodulation Therapy (PBM therapy):

PBM will be given with 940nm long infrared wavelength diode laser with following specifications Biolase Epic X Diode LASER (USFDA and CE approved) LASER Classification- IV Medium- InGaAsP Semi-Conductor Diode Wavelength- 940+10nm Maximum Output Power= 10W Pulse repetition rate= upto 20kHz Pulse duration Rate= 0.01ms- 20ms Power modes- Continuous/ Pulsed Protocol for PhotoBioModulation( PBM) therapy Protocol for PBM therapy has been made as per guidelines of the consensus statement ( Zelcha et al 2016) regarding the applications, protocols, safety, dosimetric considerations of PBM in management of side effects of chemoradiation therapy in Head and neck cancers like mucositis and fibrosis.

Protective laser wavelength specific eyewear will be used for patient, operator. The device will be used according to the manufacturer's instructions and calibration before each therapy in the trial. The surgical handpiece (diameter 0.6cm) will be used without the fibre optic tips in defocused mode and head sanitized before therapy.

Peak Power : 0.3Watts Power density: 1 Watt/cm2 Fluence: 4J/cm2 per cycle Spot size : 0.28cm2 Distance : 2mm from surface Mode: Continuous, Non- contact mode, circular motion, overlapping, in clockwise concentric manner with laser handpiece perpendicular to surface Duration of cycle : 20 seconds with interval of 30 seconds alternating with other side Cycles per sitting: Three for each side Four Sittings: Day 0,3, 7, and 15 Intraoral: Bilateral buccal mucosa will be divided arbitrarily into three zones superior, middle and inferior for equal distribution of laser energy during each cycle Extraoral :Bilateral masseter muscle will be divided into three zones superior, middle and inferior for equal distribution of laser energy during each cycle Therapeutic monitoring: Site of application of LASER will be evaluated continuously for any discomfort, signs of inflammation like redness of skin/ mucosa during therapy and during follow up. The following options will be considered during therapy Move the Handpiece relative to the affected anatomy. Defocus the energy by moving the Handpiece further away from the skin. Decrease the power setting.(considering the Fitzpatrick Skin type scale) Stop/ Defer the treatment. Patient will be interviewed to know any adverse effects they might be feeling after initiation of treatment with Laser.

Training of operators:

All the operators giving intraoral and extraoral PBM therapy will be trained in the protocol as per study before subject recruitment.

Withdrawal criteria: If any patient withdraws consent after treatment is initiated or develops any of the conditions mentioned in exclusion criteria, the patient will be withdrawn from the study.

Protocol Deviation : When/If subjects develop changes suspicious of malignancy (erosion, ulceration, induration, exophytic growth) during follow up after Usual care/PBM, they will undergo incisional biopsy to rule out malignant changes and managed as per institutional protocol for oral malignant lesions by referral to cancer center at IRCH.

Statistical Analysis: Data will be entered in an electronic data form and managed using Research Electronic Data Capture (REDcap) software. Comparison of baseline continuous variables will be compared between the two groups( A and C, B and C) using Unpaired T-test and categorical variables will be compared using Chi Squared Test or Fisher's Exact Test. The primary outcome measure- Interincisal Distance at maximum mouth opening will be compared between the two groups using Unpaired T-test and analyzed using Intention to Treat and Per Protocol Analysis. Secondary continuous outcome variables will be compared between the two groups using Unpaired T-test or Wilcoxon Rank Test as appropriate. Secondary categorical outcome variables will be compared between the two groups for two proportions/Z-test. Comparison between primary and secondary outcome variables between groups A and B will also be done using the same scheme although the sample size is not estimated for the same. Results will be presented as Difference in Means/Proportions with 95% confidence interval and p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

Subjects with symptomatic bilateral Moderate≥ 18 years of age Subjects who have had no medical, surgical or physical intervention for OSMF at least three months prior to participation in this study.

Subjects willing to participate in the study

-

Exclusion Criteria:

Subjects with any other Oral potentially malignant disorders ( Leukoplakia/ Oral lichen planus etc ) other than OSMF.

Subjects with OSMF with dysplasia in previous biopsy, suspicious lesion that requires biopsy for histopathological examination Subjects with any current / past history of any malignancies Subjects with any developmental disorders, cranio-maxillomandibular bony pathologies/ trauma, current odontogenic / maxillofacial infection or surgeries causing trismus Subjects with uncontrolled systemic diseases, psychiatric disorders o Subjects with open wounds on the sites to be exposed to LASER PBM or to EMG. Subjects with any scars, tattoos, moles, traumatic, ulcerative, pathological skin lesion on facial skin in region of masseter muscle Subjects unwilling to shave facial hair for electromyography. Subjects with history of Autoimmune diseases like Scleroderma, Dermatomyositis, oral vesiculobullous and Behçet's disease Subjects with history of any corticosteroid, immunosuppressive, anti inflammatory ,immune modulating medication in past six months Subjects with Temporomandibular Joint disorders, Cervical spondylosis muscle dystrophy or any neuromuscular disorders Pregnancy

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximal Interincisal Mouth opening (mm): | Baseline, after 1 and 3 months of PBMT
  It is described as the greatest distance between incisal edge of maxillary central incisor to the incisal edge of mandibular central incisor, when the mouth is opened as wide as possible painlessly or as the inter incisal distance plus the overbite It will be measured using Vernier calipers as described by Wood et al.

SECONDARY OUTCOMES:
Cheek Flexibility (mm): | Baseline, after 1 and 3 months of PBMT
  Cheek Flexibility (mm): Measurement of Cheek flexibility was done in accordance with the method by Mathur and Jha: Cheek flexibility = V1-V2. Two points measured at one-third the distance from the angle of the mouth on a line joining the tragus of the ear and the angle of the mouth (V2). The subject is then asked to blow his cheeks fully and the distance measured between the two points marked on the cheek (V1)
Visual Analogue Score for Pain (0-10): | Baseline, after 1 and 3 months of PBMT
  Clinical evaluation for burning sensation will be done by visual analog scale (VAS) which is a numeric rating scale of 0-10 scores, where 0 means no symptoms and 10 means severe symptoms as perceived by the individual.
Visual Analogue Score for Burning Sensation (0-10): | Baseline , after 1 and 3 months of PBMT
  Clinical evaluation for burning sensation will be done by visual analog scale (VAS) which is a numeric rating scale of 0-10 scores, where 0 means no symptoms and 10 means severe symptoms as perceived by the individual.
Electromyography evaluation of Masseter Muscle (μV): | Baseline , after1 and 3 months of PBMT
  Electromyography evaluation of Masseter Muscle (μV):
  Subjects will be instructed to maintain a natural head position shielded room to eliminate outside electrical interferences. To place the electrodes, the test, which consists of muscular palpation during simultaneous bilateral isotonic contraction, will be performed. For the masseter, electrodes will be placed between the gonion and body of the zygomatic bone. Ground electrodes will be placed on the respective mastoid process. EMG activity will be recorded at rest and maximal voluntary contraction. Time to fatigue will be recorded as time (in seconds) during which the muscles on both sides were able to perform maximum contraction until pain due to fatigue was first perceived by the patient.
Molecular characteristics of inflammatory and fibrogenic salivary cytokines (IL6, TNFα, TGFβ, CTGF) pre and post PBM therapy | Baseline, after1 and 3 of PBMT
  Four Sterile PVA ophthalmic sponges (Merocel) will be used to collect samples of oral secretion ns for four cytokine study from the oral buccal mucosa.The sponges will be pre-wet with sterile normal saline, kept in contact with the lesion/ buccal mucosa without rubbing or movement for 1 minute and then immediately stored in sterile containers at -80 °C till further analysis by ELISA.

OTHER OUTCOMES:
Maximal Interincisal Mouth opening (mm): | 6 months and 1 year after PBMT
  It is described as the greatest distance between incisal edge of maxillary central incisor to the incisal edge of mandibular central incisor, when the mouth is opened as wide as possible painlessly or as the inter incisal distance plus the overbite It will be measured using Vernier calipers as described by Wood et al.

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Gupta, MDS, FDSRCS(Edin), Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No
other researchers can contact the PI Shalini Gupta for queries about the study via email shalinigupta@hotmail.com

REFERENCES:
- [Background] Qin X, Ning Y, Zhou L, Zhu Y. Oral Submucous Fibrosis: Etiological Mechanism, Malignant Transformation, Therapeutic Approaches and Targets. Int J Mol Sci. 2023 Mar 5;24(5):4992. doi: 10.3390/ijms24054992. PMID 36902423
- [Background] More CB, Das S, Patel H, Adalja C, Kamatchi V, Venkatesh R. Proposed clinical classification for oral submucous fibrosis. Oral Oncol. 2012 Mar;48(3):200-2. doi: 10.1016/j.oraloncology.2011.10.011. Epub 2011 Nov 8. PMID 22070918
- [Background] Sukanya D, Upasana L, Deepak TA, Abhinethra MS, Choudary S. Determination of Effectiveness of Photobiomodulation in the Treatment of Oral Submucous Fibrosis. J Pharm Bioallied Sci. 2022 Jul;14(Suppl 1):S475-S478. doi: 10.4103/jpbs.jpbs_673_21. Epub 2022 Jul 13. PMID 36110778